CLINICAL TRIAL: NCT07223723
Title: A Multicenter, Open-Label, Postmarketing Surveillance Study of Tofersen (BIIB067) in Adults With Amyotrophic Lateral Sclerosis (ALS) Associated With a Mutation in the Superoxide Dismutase 1 (SOD1) Gene in China
Brief Title: A Study to Learn More About the Long-Term Safety of Tofersen (Qalsody) in Chinese Participants With SOD-1 Amyotrophic Lateral Sclerosis (ALS)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 233AS402
Record Dates: First submitted 2025-10-31; First posted 2025-11-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — tofersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tofersen 100 milligrams (mg) (Experimental): Participants will receive tofersen 100 mg by intrathecal (IT) injection as 3 loading doses once every 2 weeks (Days 1, 15, and 29), followed by 10 maintenance doses once every 4 weeks (approximately every 28 days), for a maximum total of 13 doses per participant over a 44- week treatment period.
  Interventions: Drug: Tofersen

INTERVENTIONS:
Drug: Tofersen — Administered by IT injection.
  Other Names: BIIB067, QALSODY

SUMMARY:
In this study, researchers will learn more about the safety of tofersen, also known as Qalsody®. This is a drug available for doctors to prescribe for people with a certain type of amyotrophic lateral sclerosis, also known as ALS. This type is in people who have a mutation in the superoxide dismutase 1 gene, also known as SOD-1.

This is known as a "postmarketing" study. In this kind of the study, the goal is to learn more about how a drug works after it has been approved for use in the general public. Tofersen was approved in China in September 2024. The main goal of this study is to collect long-term safety information in Chinese participants with SOD-1 ALS.

The main question researchers want to answer in this study is:

• How many participants have adverse events (AEs) and serious adverse events (SAEs)?

An AE is a health problem that may or may not be caused by a drug during the study. An AE is considered serious when it results in death, is life-threatening, causes lasting problems, or requires hospital care.

Researchers will also learn more about :

* How the body processes tofersen.
* How much tofersen is found in the cerebrospinal fluid (CSF), or the fluid that surrounds the brain and the spinal cord.

This study will be done as follows:

* Participants will be screened to check if they can join the study. The screening period will be up to 4 weeks.
* After joining the study, participants will receive the first 3 doses of 100 milligrams (mg) of tofersen about 14 days apart. This will be given through an intrathecal (IT) injection. This means it will be given into the fluid surrounding the spine.
* After that, participants will receive 10 more doses every 28 days through IT injections. Participants will have up to 13 total doses of tofersen in this study.
* Participants will have up to 15 visits to their study research center. Each participant will be in the study for up to 52 weeks (1 year).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety of tofersen in participants with SOD1-ALS in post marketing setting in China.

The secondary objective of this study is to evaluate the pharmacokinetics (PK) of tofersen in participants with SOD1-ALS in the postmarketing setting in China.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years at the time of informed consent.
* Must have diagnosis of SOD1-ALS.
* If taking riluzole, participant must be on a stable dose for ≥ 30 days prior to Day 1 and expected to remain at that dose until the final study visit.
* If taking edaravone, participant must have initiated edaravone ≥ 60 days (2 treatment cycles) prior to Day 1 and expected to remain at that dose until the final study visit, unless the Investigator determines that edaravone should be discontinued for medical reasons, in which case it may not be restarted during the study.
* All women of childbearing potential must practice effective contraception during the study.

Key Exclusion Criteria:

* Hypersensitivity to the active substance or any of the excipients of tofersen injection.
* Current or past administration of tofersen injection, in either a commercial or a clinical study setting.
* Prior or current treatment with small interfering ribonucleic acid (RNA), stem cell therapy, or gene therapy.
* Treatment with another investigational drug, biological agent, or device within 1 month or 5 half-lives of study agent, whichever is longer, prior the Baseline Visit.
* Participants who are pregnant or currently breastfeeding, and those intending to become pregnant during the study.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2027-12-16 (Estimated); Study Completion 2027-12-16 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Screening up to end of study follow-up (up to 52 weeks)

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Tofersen | Predose and at multiple timepoints postdose on Day 1
Time to Reach Maximum Plasma Concentration (Tmax) of Tofersen | Predose and at multiple timepoints postdose on Day 1
Area Under the Concentration-Time Curve (AUC) of Tofersen in Plasma | Predose and at multiple timepoints postdose on Day 1
Tofersen Cerebrospinal Fluid (CSF) Concentration | Up to 44 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Biogen
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/